CLINICAL TRIAL: NCT02272699
Title: Neoadjuvant Treatment of Nimotuzumab With Chemotherapy or Radiotherapy Versus Surgery Alone in Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Treatment of Nimotuzumab With Chemotherapy or Radiotherapy in Resectable Esophageal Squamous Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Because there are questions about adjuvant radiotherapy in this study, the clinical trial is under re-design.
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhang, Dean of the VIP-II Gastrointestinal Oncology Division of Medical Department, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCC002
Record Dates: First submitted 2014-10-11; First posted 2014-10-23 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Nimotuzumab; Neoadjuvant treatment
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — nimotuzumab; Paclitaxel; Cisplatin; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nimotuzumab with Chemotherapy (Experimental): Patients will receive neoadjuvant chemotherapy of paclitaxel and cisplatin with concurrent nimotuzumab.
  Paclitaxel 175mg per square metre on day 1 and cisplatin 30mg per square metre on day 1 and day 2 every 3 weeks for 2 cycles. Nimotuzumab 200mg per week for 6 weeks.
  After neoadjuvant treatment, patients will be evaluated by a multidisciplinary teams (MDTs) and esophagectomy will be given for patients with resectable disease.
  Interventions: Drug: Nimotuzumab; Drug: Paclitaxel; Drug: Cisplatin; Procedure: Surgery
- Nimotuzumab with radiotherapy (Experimental): Patients will receive neoadjuvant radiotherapy with concurrent nimotuzumab. Intensity-modulated radiation therapy(IMRT) of primary tumor and local lymph nodes with 95% planning target volume (PTV) of 41.4 Gy/23f. Nimotuzumab 200mg per week for 6 weeks.
  After neoadjuvant treatment, patients will be evaluated by a multidisciplinary teams (MDTs) and esophagectomy will be given for patients with resectable disease.
  Interventions: Drug: Nimotuzumab; Radiation: Radiation
- Surgery alone (Active Comparator): Patients in this group will be given esophagectomy without any neoadjuvant treatment. Adjuvant radiotherapy is permit for patients with positive lymph nodes metastasis.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab 200mg per week for 6 weeks.
  Other Names: h-R3
  Arms: Nimotuzumab with Chemotherapy; Nimotuzumab with radiotherapy
Drug: Paclitaxel — Paclitaxel 175mg per square metre on day 1, repeated every 3 weeks for 2 cycles.
  Other Names: Taxol
  Arms: Nimotuzumab with Chemotherapy
Drug: Cisplatin — Cisplatin 30mg per square metre on day 1 and day 2, repeated every 3 weeks for 2 cycles.
  Other Names: CDDP
  Arms: Nimotuzumab with Chemotherapy
Radiation: Radiation — IMRT of primary tumor and local lymph nodes with 95% PTV of 41.4 Gy/23f. Nimotuzumab 200mg per week for 6 weeks.
  Arms: Nimotuzumab with radiotherapy
Procedure: Surgery — Esophagectomy
  Arms: Nimotuzumab with Chemotherapy; Surgery alone

SUMMARY:
Esophageal cancer is one of common malignant tumors in China and esophageal squamous cell carcinoma (ESCC) is the dominant pathological type, accounting for more than 95% of all cases. One of our phase Ⅱ study introduced a combination treatment of an anti epithelial growth factor receptor (EGFR) agent, nimotuzumab, with paclitaxel and cisplatin as first-line treatment in unresectable or metastatic ESCC. The results showed that the overall response rate was 51.8% (29/56) and disease control rate was 92.9% (52/56). As a median follow-up of 24 months, the median progression-free survival for patients with metastatic disease and local advanced disease were 8.2 months and more than 23 months respectively. The overall survival for patients with metastatic disease was 13.9 months. It implied that as first-line chemotherapy, an addition of nimotuzumab to chemotherapy was a more active treatment option compared to other regimens published in previous studies. Investigations by Liang, J. and Ling, Y. also suggested that nimotuzumab in combining with radiotherapy or chemotherapy also showed anti-tumor activities and limited toxicities.

Therefore, we initiated this phase Ⅱ to Ⅲ clinical trial in which combining neoadjuvant treatments of nimotuzumab with chemotherapy or nimotuzumab with radiotherapy are compared with surgery alone for resectable stage Ⅱa to Ⅲ middle and lower thoracic esophageal squamous cell carcinoma patients. We hope to explore if these neoadjuvant combination treatments could bring survival benefit for ESCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.
* Weight loss must be less than 10% in last 6 months.
* With an expected life expectancy of ≥ 12 months
* With a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Patients must have histologically confirmed esophageal squamous cell carcinoma without prior treatments including surgery, chemotherapy, radiotherapy, and targeting treatment.
* With resectable disease of primary tumor in middle or lower thoracic esophagus and clinical stage Ⅱa-Ⅲ.
* With measurable or evaluable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Without serious system dysfunction and could tolerate chemotherapy or radiotherapy.
* Patients must have normal marrow function with a hemoglobin (HGB) of ≥90g/L, an white blood cell (WBC) counts of ≥4.0×109/L，a neutrophil count of ≥2.0×109/L, , a platelet count of ≥100×109/L, a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL), a creatinine (Cr) of ≤ 1.5 UNL, alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL.
* Patients must have normal electrocardiogram results and no history of congestive heart failure.
* Women of childbearing age should voluntarily take contraceptive measures.
* Without drug addition
* Patients must be with good compliance and agree to accept follow-up of disease progression and adverse events.

Exclusion Criteria:

* Allergic to known drug
* Patients who have received prior treatment including chemotherapy, radiotherapy and surgery.
* With unresectable disease including any T4b or M1 disease.
* Without measurable or evaluable disease.
* With history of other tumors except for those of cervical carcinoma in situ or skin basal cell carcinoma who had been completely treated and without relapse in last 5 years.
* With serious diseases such as congestive heart failure, uncontrolled myocardial infarction and arrhythmia, liver failure and renal failure.
* With neurological or psychiatric abnormalities that affect cognitive.
* Pregnant or lactated women (premenopausal women must give urine pregnancy test before enrollment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  From the date of randomization until the date of first documented relapse of disease or date of death from any cause, whichever came first. An expected average of 2 years.

SECONDARY OUTCOMES:
Overall survival | 3 years
  From the date of randomization until the date of death from any cause. An expected average of 3 years.
Pathological complete response of neoadjuvant treatment | 4 months
  From the date of randomization until the date of pathological diagnosis is reported after esophagectomy. An expected average of 4 months.
The R0 resection rate | 3 months
  From the date of randomization to one week after the surgical resection of tumor (esophagectomy). An expected average of 3 months.
Numbers of adverse events and the degree of each adverse events according to the NCI CTCAE 4.0 criteria. | 6 months
  From the date of randomization to 3 months after esophagectomy. An expected average of 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhang, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital & Peking University Cancer Hospital, Beijing, Beijing Municipality, China